CLINICAL TRIAL: NCT05303922
Title: Dual-Energy Computed Tomography (DECT) in Acute Neck Infections: Comparison With Magnetic Resonance Imaging (MRI) (ANI-DECT)
Brief Title: Dual-Energy Computed Tomography (DECT) in Acute Neck Infections: Comparison With Magnetic Resonance Imaging (MRI)
Acronym: ANI-DECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Jussi Hirvonen, Radiologist, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T257/2021
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Neck Abscess
Keywords: Computed tomography; Magnetic resonance imaging

STUDY DESIGN:
Intervention Model Description: Each patient will be scanned with both DECT and MRI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DECT and MRI (Experimental): Patients will be scanned with both DECT and MRI.
  Interventions: Diagnostic Test: Dual-energy CT; Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: Dual-energy CT — Dual-energy CT
Diagnostic Test: MRI — MRI

SUMMARY:
The purpose of this prospective study is to compare MRI and DECT in imaging acute neck infection. 50 patients suspected for neck infection will undergo both modalities, which will then be compared in terms of depiction of edema, conspicuity of inflammation, and characterization and number of abscesses. We hypothesize that DECT will have diagnostic performance comparable to that of MRI, and superior to that of traditional single-energy CT. This study will yield important new information about the performance of DECT, a novel and rapid method for emergency imaging.

DETAILED DESCRIPTION:
Deep neck infections present challenges even in modern medicine, due to complex anatomy and potentially lethal complications. True extent of the infection is difficult to assess clinically. Therefore, medical imaging is useful in determining the exact location and extent of disease. In suspected neck infection, computed tomography (CT) has traditionally been the first-line imaging method. However, magnetic resonance imaging (MRI) provides excellent soft-tissue characterization surpassing that of CT in the initial evaluation of neck infections. Previous studies have shown than MRI is superior to CT in terms of lesion conspicuity and number of affected spaces in neck infections. As an alternative to MRI, dual-energy CT (DECT) could offer improved soft tissue sensitivity compared with traditional single-energy CT. DECT refers to CT imaging carried out with two kinds of spectra of x-ray. In this prospective comparative study, we will recruit emergency patients with suspected neck infection. Neck MRI will be completed as part of standard clinical care, and DECT as part of this research study. After study completion, DECT and MRI will be compared by neuroradiologists, both modalities at separate occasions, blinded to the clinical information and diagnosis as well to the result of the other modality. Clinical care will be based on MRI as is usual practise. Surgical findings will be considered gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Suspicion of acute neck infection as deemed by the referring physician

Exclusion Criteria:

* History of a serious adverse reaction to intravenous iodine- or gadolinium-based contrast agent
* Severe kidney dysfunction (eGFR < 30 mL/min/1.73m2)
* Foreign metallic objects incompatible with MRI in the body
* Inability to give informed consent, as deemed by study physician
* Inability to follow study instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1 day
  Diagnostic accuracy relative to clinical reference standard (clinical diagnosis or surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Hirvonen, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No